CLINICAL TRIAL: NCT02772848
Title: A Prospective Collection of Peripheral Blood Specimens to Study Fertility in Healthy, Premenopausal Women
Brief Title: Fertility in Healthy Premenopausal Women
Status: Completed | Type: Observational
Sponsor: Fujirebio Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FDI-81
Record Dates: First submitted 2016-04-19; First posted 2016-05-16 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-04

CONDITIONS: Fertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The study objectives are described below:

1. Obtain serum specimens collected for one ovulatory cycle or a maximum of 33 days, but not to exceed a total of 550 ml of whole blood per subject from a minimum of 60 healthy, premenopausal subjects. Specimens will be used to determine a reference range for estradiol, FSH, LH, and progesterone assays, used as an aid in the assessment of fertility in adult, premenopausal women.
2. To store any remaining specimens for use in future assay development and to evaluate as yet undetermined assays for the development of IVDs, including additional estradiol, FSH, LH, and progesterone assays.

DETAILED DESCRIPTION:
The purpose of this study is to obtain sufficient specimens and correlating clinical data from a well-controlled prospective clinical trial collecting specimens from healthy, premenopausal subjects to support domestic and international regulatory submissions on fertility biomarker assays, and to establish a collection of specimens that will support future assay discovery and validation efforts.

ELIGIBILITY:
Inclusion Criteria:

* Females, age ≥ 21 years
* Premenopausal (defined as a woman that has had at least one menstrual cycle in the last 365 days).
* A minimum weight of 110 lbs
* The subject is not anemic (Hemoglobin ≥ 12.5 g/dL)
* Willing to provide a daily blood draw for one ovulatory cycle or a maximum of 33 days
* Able to understand and willing to provide informed consent.

Exclusion Criteria:

* Males
* Females, age <21 years
* Weighing < 110 lbs
* Anemic (Hemoglobin < 12.5 g/dL)
* History of bilateral oophorectomy
* Females taking any form of hormonal birth control including:

  * Oral contraceptive pill (combined or progestin-only) within five days enrollment.
  * Contraceptive patch (such as Ortho Evra®) within seven days of enrollment.
  * Vaginal contraceptive ring (such as NuvaRing™) within 21 days of enrollment.
  * Contraceptive injection (such as Depo-Provera®) within 90 days of enrollment.
  * Intra-uterine system (IUS) within 90 days of enrollment. An intra-uterine device (IUD) made of copper does not exclude the patient from participating in this study.
  * Subdermal contraceptive implants (such as Nexplanon®) within 90 days of enrollment.
  * Emergency contraceptive within 30 days of enrollment.
* Women in menopause (defined as the end of menstrual cycles or at least more than 365 days since the last menstrual cycle)
* Amenorrhea except for women that continue to ovulate as documented in a physician note available to the enrolling center.
* Has a current diagnosis of any clinically significant cardiac, respiratory, neurological, immunological, hematological, liver disease, renal disease, gastrointestinal (GI) disorder, including any history of hyper- or hypothyroid, peptic or gastric ulcers or GI bleeding, or any other condition which, in the opinion of the investigator, would deem the subject unhealthy and therefore, ineligible.
* Has a history of any clinically significant cardiac, respiratory, neurological, immunological, hematological, liver disease, renal disease, gastrointestinal (GI) disorder, including any history of hyper- or hypothyroid, peptic or gastric ulcers or GI bleeding, or any other condition which, in the opinion of the investigator, is unstable at the time of enrollment.
* Is receiving systemic chemotherapy or radiation treatment, has an active malignancy of any type, or has been diagnosed with cancer within 5 years before screening other than basal or squamous cell skin cancers or in-situ cervical cancer.
* History of seizures
* Diagnosed with an infectious disease including any sexually transmitted diseases.
* Diagnosed with HIV/AIDS or ever tested positive for HIV.
* History of hepatitis
* Subject that has had sexual contact with a person who has hepatitis within the last 12 months.
* Pregnancy, lactation or actively seeking to conceive (trying to become pregnant).
* Unable to provide informed consent.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A minimum of 60 subjects will be enrolled in this study. Healthy, premenopausal women greater than or equal to 21 years of age having donated a serial blood collection throughout a single ovulation cycle or a maximum of 33 days will be eligible.
  Each site or mobile center will evaluate and select patients for enrollment using the inclusion and exclusion criteria listed below. Study subjects should be selected from all available patients at the site or mobile center. Each patient may be entered into the study only once. Subject enrollment and/or Day 1 blood draw is not associated with a specific time point in the ovulatory cycle.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Measurement of fertility hormone levels in 60 + healthy premenopausal women | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Diana Dickson, Study Director — Fujirebio Diagnostics, Inc.
Locations (2):
- United States (2):
  - Vita Pharma, Hialeah, Florida
  - American Blood Bank, Inc., Miami, Florida

IPD SHARING:
Plan to Share IPD: No